CLINICAL TRIAL: NCT02846311
Title: Prospective Evaluation of the Alere i Influenza A&B Nucleic Acid Amplification Versus Xpert Flu/RSV
Brief Title: Evaluation of the Alere i Influenza A&B Nucleic Acid Amplification Versus Xpert Flu/RSV
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Test iFluA&B
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2016-07

CONDITIONS: Influenza
Keywords: test; winter; season
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group with support that will be usually performed: During the first phase ("before"), the assumption will be that usually achieved.
  The doctor continues to support according to information it has and according to good practice and service protocols.
- Group with a flu test: During the second phase ("after"), a flu test is routinely performed within the home emergency department by the doctor who supports the patient.
  The doctor continues to support according to information it has and according to good practice and service protocols.
  Interventions: Device: Flu Test

INTERVENTIONS:
Device: Flu Test
  Groups: Group with a flu test

SUMMARY:
The rapid and accurate detection of influenza virus in respiratory specimens is required for optimal management of patients with acute respiratory infections. Because of the variability of the symptoms and the numerous other causes of influenza-like illness, the diagnosis of influenza cannot be made on the basis of clinical criteria alone. Thus, rapid influenza diagnostic tests have been developed such as the Alere i Influenza A&B isothermal nucleic acid assay. Investigators prospectively evaluated the performance of the Alere i Influenza A&B assay in comparison with the routine Xpert Flu/RSV assay.

DETAILED DESCRIPTION:
Main objective / secondary:

It appears that so far the weight of the influenza disease, the limits of clinical diagnosis and validity of rapid diagnostic methods to emergencies are well studied and validated. However the potential organizational and economic benefit in emergency care services remains little known and rarely evaluated.

The significant improvement in diagnostic response time he has a real beneficial impact for the patient? For the organization of the emergency? Investigators propose to study the impact of the implementation of rapid diagnostic solution by molecular biology of influenza directly available in an adult emergency department, from a cohort of patients consulting in connection a flu-like illness. Investigators wish in particular to highlight the organizational and economic impact.

Methodology :

DESIGN:

Study single-center, prospective, descriptive, observational, type "before / after".

Unable to reasonably perform a prospective randomized study due to the constraints for patients and for the service and means that it would be necessary to deploy in this case (CRA ... PHRC), Methodology :

DESIGN:

Study single-center, prospective, descriptive, observational, type "before / after".

Unable to reasonably perform a prospective randomized study due to the constraints for patients and for the service and means that it would be necessary to deploy in this case (CRA ... PHRC), we are moving more towards a comparison study before / after between February and April.

Time study Total study duration: 3 months Inclusion period: 3 months (February 2016- April 2016)

Acquisition of data:

Data Observing Notebook (CRF or "Case Report Form") are disclosed in the notes accompanying this document and will be collected aur an Excel spreadsheet Statistical analysis ( For each subject will be awarded an identifier (original name and surname - year of birth) and the data will be entered on a computer file which will be sent to the statistician in charge of analyzing the GHPSJ site. There will be no exchange of personal data for this study is single center on the site GHPSJ.

Development of the study:

The patient presents to the Emergency Home Service for a "flu syndrome". During the first phase ( "before"), the assumption will be that usually achieved.

During the second phase ( "after"), a flu test is routinely performed within the home emergency department by the doctor who supports the patient.

In both cases, the doctor continues to support according to information it has and according to good practice and service protocols.

A case report form (CRF or Case Report Form) is completed for each patient included in the study. This report forms includes a questionnaire that collects anonymous demographic information (patient age and sex) and clinical data. The CRF also includes the results of the rapid test for influenza. These notebooks anonymous comments are seized by the Home Emergency Service on a type of database "Access" (which will then be completed by the results of the rapid test. If positive, strain characterization will be clarified.

Number of patients recruited (justification) and duration of participation for each patient:

Not applicable as observational study are moving more towards a comparison study before / after between February and April.

Time study Total study duration: 3 months Inclusion period: 3 months (February 2016- April 2016)

ELIGIBILITY:
Inclusion Criteria:

1. Respiratory Symptoms include cough, dyspnea and / or
2. General symptoms: headache, myalgia, asthenia, anorexia ... and / or
3. Acute fever above 38 ° C
4. Patient consent.

Exclusion Criteria:

* Major cognitive disorders
* Patient under guardianship
* Patient refusing to consent to research
* Duplicate (patients who have had laboratory diagnosis of influenza in previous 7 days)
* Patient not receiving social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (> 18 years) consultant to the ER for influenza-like illness involving
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Assessment of change of the Length of stay in the emergency service | Day 1
  Will be assessed with patients of the firt group (phase 1) and the second one (With Flu Test)
Assessment of change of Hospitalization rates | Day 1
  Will be assessed with patients of the firt group (phase 1) and the second one (With Flu Test)

SECONDARY OUTCOMES:
Assessments of change of antibiotic treatment Costs | Day1
  Will be assessed with patients of the firt group (phase 1) and the second one (With Flu Test)

CONTACTS AND LOCATIONS:
Overall Officials: TRABATTONI Eloïse, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France